CLINICAL TRIAL: NCT02392312
Title: Safety and Efficacy of Individual Batches of ATG-F in Kidney Transplant Recipients: Multicentre, Prospective, Observational Study
Brief Title: Observational Study to Evaluate the Safety and Efficacy of ATG-F on Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ATG-MA-ACN001
Record Dates: First submitted 2015-03-13; First posted 2015-03-18 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-01

CONDITIONS: Kidney Transplant Recipients
Keywords: kidney transplant; ATG-F

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATF-Fresenius S: intravenous
  Interventions: Drug: ATF-Fresenius S

INTERVENTIONS:
Drug: ATF-Fresenius S — intravenous

SUMMARY:
A multicenter, prospective, observational study to evaluate the safety and efficacy of individual batches of ATG-F in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* ATG-F administration to prophylaxis rejection in kidney transplantation recipient.
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study is obtained.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients.).
* Subjects with bacterial, viral, mycotic or parasitic infections, which are not under adequate therapeutic control.
* Solid organ transplant subjects with severe thrombocytopenia, i.e. less than 50,000 platelets/µl because ATG-F may enhance thrombocytopenia and thus increase the risk of hemorrhage.
* Current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix that has been treated successfully.
* Subject is receiving a Human Leukocyte Antibody (HLA) identical living donor organ.
* Subject is unlikely to comply with the visits scheduled in the protocol in the opinion of investigator or has a history of non-compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Governmental Hospital
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse event | up to 3 months post-transplantation

SECONDARY OUTCOMES:
Clinical diagnosis of acute rejection | up to 3 months post-transplantation
Renal function: serum creatinine | at month 1 and month 3
Incidence of delayed graft function (DGF) | up to 3 months post-transplantation
Patient and graft survival | up to 3 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma China, Inc.
Locations (25):
- China (25):
  - Site: CN00004, Baotou
  - Site: CN00011, Beijing
  - Site: CN00012, Beijing
  - Site: CN00013, Beijing
  - Site: CN00016, Changchun
  - Site: CN00002, Chengdu
  - Site: CN00003, Chongqing
  - Site: CN00018, Fuzhou
  - Site: CN00023, Guangzhou
  - Site: CN00021, Haikou
  - Site: CN00022, Haikou
  - Site: CN00019, Hangzhou
  - Site: CN00020, Hangzhou
  - Site: CN00006, Jinan
  - Site: CN00017, Jinan
  - Site: CN00028, Kunming
  - Site: CN00030, Nanchang
  - Site: CN00015, Qingdao
  - Site: CN00010, Shiyan
  - Site: CN00014, Taiyuan
  - Site: CN00005, Tianjin
  - Site: CN00031, Ürümqi
  - Site: CN00001, Xi'an
  - Site: CN00033, Yantai
  - Site: CN00007, Zhengzhou

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.